CLINICAL TRIAL: NCT00808977
Title: A Double-blind, Randomised, Placebo and Mesalazine Controlled Phase II Study to Explore the Safety and Activity of Dersalazine in Patients With Mild to Moderate Active Colitis
Brief Title: A Phase II Study to Explore the Safety and Activity of Dersalazine in Patients With Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palau Pharma S.L.U. (Industry)
Responsible Party: Caridad Pontes / Head Clinical Research, Palau Pharma S.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR-IBD-1-08; EudraCT 2008-004610-27 (Registry Identifier: Eudra CT)
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — dersalazine; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dersalazine (Experimental)
  Interventions: Drug: Dersalazine sodium
- Mesalazine (Active Comparator)
  Interventions: Drug: Mesalazine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dersalazine sodium — Dersalazine sodium 2400 mg daily
  Arms: Dersalazine
Drug: Mesalazine — Mesalazine 2400 mg daily
  Arms: Mesalazine
Drug: Placebo — Placebo matching active and experimental treatments
  Arms: Placebo

SUMMARY:
The purpose of the study is to obtain a first clinical assessment of the safety of dersalazine sodium in ulcerative colitis patients with mild to moderate disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 inclusive
* Male, non-child-bearing female or fertile female with appropriate contraception.
* Mild to moderate confirmed active ulcerative colitis
* Able and willing to give informed consent

Exclusion Criteria:

* Colitis of other cause
* Pregnancy, inadequate contraception for fertile female patients
* Liver or kidney disease, unstable cardiovascular disease, coagulation disorder.
* Other significant medical condition that preclude participation at investigator criteria
* Allergy or hypersensitivity to salicylates
* Previous or concomitant treatment for ulcerative colitis interfering with safety or activity assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with AEs of severe intensity or AEs leading to treatment withdrawal | 7, 14, 21, 28, 56 days

SECONDARY OUTCOMES:
Mayo index | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Julian Panés, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (22):
- Belgium (2):
  - Investigational site 11, Kortrijk
  - Investigational site 1, Leuven
- Hungary (5):
  - Investigational site 12, Budapest
  - Investigational site 10, Eger
  - Investigational site 9, Miskolc
  - Investigational site 8, Székesfehérvár
  - Investigational site 7, Vác
- Slovakia (5):
  - Investigational site 18, Košice
  - Investigational site 20, Košice
  - Investigational site 16, Malacky
  - Investigational site 17, Nové Zámky
  - Investigational site 19, Rožňava
- Spain (10):
  - Investigational site 2, Badalona
  - Investigational site 15, Barcelona
  - Investigational site 3, Barcelona
  - Investigational site 5, Barcelona
  - Investigational site 21, Cadiz
  - Investigational site 6, Córdoba
  - Investigational site 22, Madrid
  - Investigational site 14, Sabadell
  - Investigational site 13, Terrassa
  - Investigational site 4, Terrassa

REFERENCES:
- [Derived] Pontes C, Vives R, Torres F, Panes J. Safety and activity of dersalazine sodium in patients with mild-to-moderate active colitis: double-blind randomized proof of concept study. Inflamm Bowel Dis. 2014 Nov;20(11):2004-12. doi: 10.1097/MIB.0000000000000166. PMID 25192498
- [Derived] Roman J, Planell N, Lozano JJ, Aceituno M, Esteller M, Pontes C, Balsa D, Merlos M, Panes J, Salas A. Evaluation of responsive gene expression as a sensitive and specific biomarker in patients with ulcerative colitis. Inflamm Bowel Dis. 2013 Feb;19(2):221-9. doi: 10.1002/ibd.23020. PMID 22605655